CLINICAL TRIAL: NCT01369979
Title: Hepatic Glucose Metabolism Measured by FDG PET/CT in Patients With Liver Disease and Healthy Subjects
Brief Title: Hepatic Sugar Metabolism Measured by PET/CT in Patients and Healthy Subjects
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 20100284
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Liver Cirrhosis
Keywords: Lumped constant; FDG; PET
MeSH Terms: conditions — Liver Cirrhosis | interventions — Cooking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma for measuring levels of ICG, insulin, c.peptide, FFA, glucagon,and 3H-glucose.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with chronic liver disease: Inclusion criteria
  * Age between 40 and 70 years
  * BMI between 20 and 26
  Exclusion Criteria
  * Diabetes mellitus
  * Glucose intolerance
  * Medical treatment of portal hypertension
  * People who have undergone surgery for obesity
  * Pregnancy
  Interventions: Procedure: Liver vein catheter
- Healthy subjects: Inclusion criteria
  * Age between 40 and 70 years
  * BMI between 20 and 26
  Exclusion Criteria
  * Diabetes mellitus
  * Glucose intolerance
  * Medical treatment of portal hypertension
  * People who have undergone surgery for obesity
  * Pregnancy
  Interventions: Procedure: Liver vein catheter

INTERVENTIONS:
Procedure: Liver vein catheter — Liver vein catheter is placed in the heptic vein via the femoral vein, using fluoroscpoy as guidance.
  Other Names: Cook, Torcon NB Advantage Catheter

SUMMARY:
The investigators wish to determine the lumped constant (LC), which is a correction factor necessary for converting measurements of hepatic FDG metabolism (measured by PET) to those of regular glucose in patients with cirrhosis and healthy subjects.

Working hypothesis

* LC for FDG in liver tissue is not significantly different from unity in healthy subjects
* LC for FDG in liver disease is significantly different from LC in healthy liver
* Insulin changes the LC for FDG in liver tissue, but not by the same factor in liver disease and healthy subjects.

DETAILED DESCRIPTION:
The LC for FDG is determined in 8 patients with liver disease and 8 healthy volunteers with and without glucose-clamp on two different days at 3-5 week intervals. The individual order of the two examinations will be randomized. The subjects fast overnight before the examination but are allowed to drink water and take usual medication.

When arriving at the PET centre, venflons are placed in a cubital vein in both arms and an ICG infusion is started in one of them. On the day with the glucose-clamp, an infusion of insulin and glucose is started in the second venflon. Next, an artflon is placed in one radial artery and a lever vein catheteter is placed via an introducer catheter in the left femoral vein under sterile conditions and local anesthetic (Lidocaine). The position of the liver vein catheter is checked with fluoroscopy.

On each experimental day, a bolus of 200 MBq FDG + 25 μCi [3H] glucose (diluted with saline up to 10 ml) is given intravenously at the start of a 60-min PET scan of the liver. Blood samples from a peripheral artery and a liver vein are collected for determination of blood concentrations of FDG and [3H]glucose at appropriate intervals.

In the experiment with glucose-clamp, an intravenous infusion of insulin (0.6 mU/kg/min) is given and blood glucose is measured every 10 min and kept constant at around 5 mM by infusing 20% glucose (infusion rate adjusted according to blood glucose).

During each study, the hepatic blood flow rate is measured by giving an intravenous infusion of indocyanine green (ICG) and collecting arterial and liver vein blood samples (Fick's principle).

Blood samples are analyzed for concentrations of FDG (gammacounter), [3H]glucose (liquid-scintillation counter), glucose (enzymatic assay) and ICG (spectrophotometric).

When the experiment is finished, all infusions are terminated and the liver vein catheter is removed and hemostasis ensured by manual compression (10 minutes) and bed rest for 30 minutes before the subject is allowed to stand. The artflon is then removed and hemostasis ensured by manual compression (10 minutes). Finally, the venflons are removed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 70 years
* BMI between 20 and 26

Exclusion Criteria:

* Diabetes mellitus
* Glucose intolerance
* Medical treatment of portal hypertension
* People who have underwent surgery for obesity
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited via 2 newspapers: Århus Onsdag and Århus Stiftstidende, and so will be based in the area these newspapers are distributed in.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sørensen, MD PhD, Principal Investigator — Aarhus University Hospital, PET-centre
Locations (1):
- Aarhus University Hospital, PET-centre, Aarhus C, Denmark